CLINICAL TRIAL: NCT05497765
Title: Effects of Compound Silymarin on Biomarkers of Lipid Metabolism and Inflammation in Patients With Non-alcoholic Fatty Liver Disease: A Randomized Controlled Double-blind Trial
Brief Title: An Intervention Study of Compound Silymarin in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Honghui Guo, Professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDMUSPH001
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic fatty liver disease; Silymarin; Inflammation; Lipid metabolism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammation | interventions — Silybin; schizandrin; dan-shen root extract

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compound silymarin (Experimental): Dietary supplement: 4 tablets of compound silymarin twice a day for 12 weeks The active ingredient in each tablet: 81.6 mg of silibinin, mixed power of pueraria, schisandra and salvia miltiorrhiza
  Interventions: Dietary Supplement: Silibinin extract, mixed power of pueraria, schisandra and salvia miltiorrhiza
- Silymarin (Active Comparator): Dietary supplement: 4 tablets of silymarin twice a day for 12 weeks The active ingredient in each tablet: 81.6 mg of silibinin
  Interventions: Dietary Supplement: Silibinin extract
- Placebo (Placebo Comparator): Dietary supplement: 4 tablet of placebo twice a day for 12 weeks Placebo Composition: corn dextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Silibinin extract, mixed power of pueraria, schisandra and salvia miltiorrhiza — Take 4 tablets with warm water twice a day
  Arms: Compound silymarin
Dietary Supplement: Silibinin extract — Take 4 tablets with warm water twice a day
  Arms: Silymarin
Dietary Supplement: Placebo — Take 4 tablets with warm water twice a day
  Arms: Placebo

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has become the most prevalent liver disorder in China. The aim of this project is to evaluate the effects of compound silymarin on biomarkers of lipid metabolism and inflammation in the patients with NAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) has become the most prevalent liver disorder in China but still has no exact therapy for this disease instead of improving our diet and enhancing physical activity. Silymarin is a mixture of flavonoids extracted from seeds of Silybum marianum or milk thistle, and its major active compound is silibinin. Because of its antioxidant, anti-inflammatory and antifibrotic power, silymarin has important biological effects in NAFLD. Furthermore, some traditional liver protective Chinese medicines are also helpful in controlling the progression of NAFLD, such as pueraria, schisandra and salvia miltiorrhiza. At present, there are few reports on the combination of silymarin and these traditional Chinese medicines in the treatment of NAFLD. This study aims to test the effect of compound silymarin on laboratory markers and clinical evolution of patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Subject's BMI is ≥ 22.0 kg/m2 and < 33.0 kg/m2;
* Subject is diagnosed with NAFLD according to the Chinese Non-alcoholic fatty liver disease prevention guide 2018;
* A mildly elevated of ALT level (≥ 30 U/L for male, ≥ 19 U/L for female) or an AST/ALT ratio < 1.0;
* Must be able to swallow tablets.

Exclusion Criteria:

* ≥ 30 grams of alcohol/day for male and ≥ 20 grams of alcohol/day for female;
* Patients with certain hepatic diseases such as gallstones, hepatitis C, autoimmune hepatitis, and hepatolenticular degeneration which can lead to fatty liver disease;
* Be taking medicines or supplements that would influence the liver function, lipid metabolism;
* Patients with total parenteral nutrition, inflammatory bowel disease, celiac disease, hypothyroidism, Cushing syndrome, Mauriac syndrome, etc;
* Patients with hereditary diseases, coronary heart disease, mental disorder, cancer, cirrhosis and renal disease;
* Body weight change are more than 10% in previous 3 months;
* Patients who have participated in or are participating in other clinical trials within 3 months of their first administration of the study product;
* Subjects are allergic to the ingredients in the test or control samples;
* Woman who is pregnant or breastfeeding;
* Subjects cannot meet the requirements of compliance in the pre-experiment period;
* Subjects who fail to sign the informed consent forms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Liver enzymes | Change from baseline ALT and AST at 12 weeks
  Serum activities of alanine transaminase (ALT) and aspartate transaminase (AST)
Lipid profile | Change from baseline lipid profile at 12 weeks
  Serum levels of total cholesterol (TC), triglyceride (TG), high density lipoprotein-cholesterol (HDL-C) and low density lipoprotein-cholesterol (LDL-C)

SECONDARY OUTCOMES:
T-Lymphocytes' composition | Change from baseline T-Lymphocytes' composition at 12 weeks
  Changes of T-Lymphocytes' composition in peripheral blood
Bile acid metabolism | Change from baseline composition of serum and fecal bile acids at 12 weeks
  Composition of serum and fecal bile acids

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, School of Public Health, Guangdong Medical University, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghemo A, Alekseeva OP, Angelico F, Bakulin IG, Bakulina NV, Bordin D, Bueverov AO, Drapkina OM, Gillessen A, Kagarmanova EM, Korochanskaya NV, Kucheryavii UA, Lazebnik LB, Livzan MA, Maev IV, Martynov AI, Osipenko MF, Sas EI, Starodubova A, Uspensky YP, Vinnitskaya EV, Yakovenko EP, Yakovlev AA. Role of silymarin as antioxidant in clinical management of chronic liver diseases: a narrative review. Ann Med. 2022 Dec;54(1):1548-1560. doi: 10.1080/07853890.2022.2069854. PMID 35635048
- [Background] Malik A, Nadeem M, Malik MI. Efficacy of elafibranor in patients with liver abnormalities especially non-alcoholic steatohepatitis: a systematic review and meta-analysis. Clin J Gastroenterol. 2021 Dec;14(6):1579-1586. doi: 10.1007/s12328-021-01491-7. Epub 2021 Aug 9. PMID 34370218
- [Background] Kalopitas G, Antza C, Doundoulakis I, Siargkas A, Kouroumalis E, Germanidis G, Samara M, Chourdakis M. Impact of Silymarin in individuals with nonalcoholic fatty liver disease: A systematic review and meta-analysis. Nutrition. 2021 Mar;83:111092. doi: 10.1016/j.nut.2020.111092. Epub 2020 Nov 25. PMID 33418491
- [Background] Navarro VJ, Belle SH, D'Amato M, Adfhal N, Brunt EM, Fried MW, Reddy KR, Wahed AS, Harrison S; Silymarin in NASH and C Hepatitis (SyNCH) Study Group. Silymarin in non-cirrhotics with non-alcoholic steatohepatitis: A randomized, double-blind, placebo controlled trial. PLoS One. 2019 Sep 19;14(9):e0221683. doi: 10.1371/journal.pone.0221683. eCollection 2019. PMID 31536511
- [Background] Zhong S, Fan Y, Yan Q, Fan X, Wu B, Han Y, Zhang Y, Chen Y, Zhang H, Niu J. The therapeutic effect of silymarin in the treatment of nonalcoholic fatty disease: A meta-analysis (PRISMA) of randomized control trials. Medicine (Baltimore). 2017 Dec;96(49):e9061. doi: 10.1097/MD.0000000000009061. PMID 29245314
- [Background] Wah Kheong C, Nik Mustapha NR, Mahadeva S. A Randomized Trial of Silymarin for the Treatment of Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1940-1949.e8. doi: 10.1016/j.cgh.2017.04.016. Epub 2017 Apr 15. PMID 28419855